CLINICAL TRIAL: NCT03615612
Title: Investigation of the Accuracy of a Low-cost, Portable, Autorefractor to Provide Well-tolerated Eyeglass Prescriptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: PlenOptika, Inc. (Industry); Aravind Eye Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00157754
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OR Eyeglasses, then SR (Other): Objective Refraction (OR) Eyeglasses, then Subjective Refraction (SR)
  Interventions: Other: QuickSee refractive error assessment + glasses
- SR Eyeglasses, then OR (Other): Subjective Refraction (SR) Eyeglasses, then Objective Refraction (OR)
  Interventions: Other: QuickSee refractive error assessment + glasses

INTERVENTIONS:
Other: QuickSee refractive error assessment + glasses — QuickSee refractive error assessment + glasses

SUMMARY:
At the Aravind Eye Hospital (AEH) in Madurai, India, patients ages 18-40 receiving treatment for refractive error who choose to enroll in the study will be evaluated using subjective refraction and objective refraction, by way of the QuickSee autorefractor. Patients will then be randomized into one of two treatment plans: receive glasses from objective measure first then subjective measure second, and vice versa. After one week of wearing the first pair of glasses, patient preferences are assessed, and glasses are switched. After a week of wearing the second pair of glasses from the alternate measurement method, patient preferences are again assessed. Patients may then decide which pair patient like best. This is a double blind, case-crossover clinical trial.

ELIGIBILITY:
Inclusion Criteria: Participants-

1. who visit a Vision Center for their eye check-up
2. who are aged between 18 years and 40 years

Exclusion Criteria: Participants-

1. whose refractive error is not within the detection range of the QuickSee device: -10 to +10 D
2. who have a cylindrical power greater than 3 D
3. who have to travel long distances (beyond 10kms) to the hospital
4. who choose to buy spectacles that are priced more than Rs. 2000/- per pair
5. who have speech or hearing impairment
6. who do not speak the local language, Tamil
7. who do not want to purchase spectacles from AEH

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Patient Preference | 2 years
  Patients are asked the question "Which eyeglasses did you prefer?". Patient response is then recorded.

CONTACTS AND LOCATIONS:
Overall Officials: David Friedman, MD, MPH, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months
Access Criteria: PlenOptika, Aravind Eye Hospital, Johns Hopkins